CLINICAL TRIAL: NCT03132506
Title: E-Health Portal for Individualized Treatment Monitoring and Patient Engagement in Oncology Research Focused on Capture of Patient Reported Outcomes with Within PRAEGNANT Study Network
Brief Title: E-Health Portal for Individualized Treatment Monitoring and Patient Engagement in Oncology Research
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: National Center for Tumor Diseases (NCT), University Hospital Heidelberg, Germany (Unknown); Department of Gynecology and Obstetrics, University Hospital Heidelberg, Germany (Unknown); Department of Gynecology and Obstetrics, University Hospital Erlangen, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pepper
Record Dates: First submitted 2017-04-12; First posted 2017-04-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- paper-based patient-reported-outcomes
  Interventions: Other: patient-reported-outcomes
- on web-based patient-reported-outcomes
  Interventions: Other: patient-reported-outcomes

INTERVENTIONS:
Other: patient-reported-outcomes — Explorative pilot study combining collected data from the PRAEGNANT study on paper-based patient-reported-outcomes with additional collected data on web-based patient-reported-outcomes

SUMMARY:
Evaluation of patient acceptance and characterization of response behaviour for web-based compared with respective paperbacked patient reported outcomes.

DETAILED DESCRIPTION:
Paperbacked pPRO data from up to a total of 100 patients from the cohort of PRAEGNANT are planned to be included in the Pepper I PRO study. Additionally 200 patients will be recruited in the web based ePRO cohort. The study duration per patient is at least 8 weeks. In cases of stable disease the study duration can be extended to up to 6 months with monthly PRO assessments, according to the attached visit matrix, taking approximately 20 minutes per visit.

The documentation at baseline should be performed during clinical routine with trained study personnel followed by remote self-reporting to minimize the patient effort. Pepper I will be conducted as sub-protocol of the PRAEGNANT trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in PRAEGNANT
* Women aged ≥18 years
* Patients with the diagnosis metastasized breast cancer undergoing any form of systemic therapy
* Patients who are willing and able to sign the informed consent form
* Patients with therapy change

Exclusion Criteria:

* Patients who are not eligible for observation due to severe comorbidities or unavailability according to the treating physician
* Patients who are not able to handle a tablet computer or are unable to write
* Patients who are not able to understand the nature and extent of the trial and the procedures require

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population for the paperbased PRO capture is part of the PRAEGNANT study population and shall comprize 100 patients, we aim to collect additional web based ePRO datasets for 200 patients
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
QLQ-C30 questionnaire for baseline | 8 weeks
  Overall patient completion rate in the paperbacked questionnaire and the web-tool, respectively

SECONDARY OUTCOMES:
All other questionnaires for baseline and follow up time points. | Baseline, 8 weeks
  Overall patient completion rate in the paperbacked questionnaire and the web-tool, respectively,
Influence factors for the completion rates | 8 weeks
  age
Influence factors for the completion rates | 8 weeks
  line of treatment
Influence factors for the completion rates | 8 weeks
  treatment
Influence factors for the completion rates | 8 weeks
  technical skills
Influence factors for the completion rates | 8 weeks
  patient's satisfaction
Adverse events-1 | 8 weeks
  The date of clinical diagnosis of AE compared with the date of early AE onset
Adverse events-2 | 8 weeks
  Consistency of AE documentation ePRO and clinician based
Patient satisfaction | baseline, 4 weeks, 8 weeks
  at baseline, after 4 weeks and after 8 weeks
Health related quality of life (HRQL) assessements -1 | baseline, 4 weeks, 8 weeks
  EORTC QLQ C-30
Health related quality of life (HRQL) assessements -1 | baseline, 4 weeks, 8 weeks
  BR23
Health related quality of life (HRQL) assessements -1 | baseline, 4 weeks, 8 weeks
  NCCN distress thermometer,
Health related quality of life (HRQL) assessements -1 | baseline, 4 weeks, 8 weeks
  EQ-VAS
Health related quality of life (HRQL) assessements -1 | baseline, 4 weeks, 8 weeks
  PHQ-9
Health related quality of life (HRQL) assessements -2 | baseline, 8 weeks
  The HRQL assessements EQ-5D-5L measured at baseline and weekly (8 weeks)
Health related quality of life (HRQL) assessements -2 | baseline, 8 weeks
  The HRQL assessements PROCTCAE Endocrine measured at baseline and weekly (8 weeks)
Health related quality of life (HRQL) assessements -2 | baseline, 8 weeks
  The HRQL assessements PROCTCAE taxane measured at baseline and weekly (8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallwiener M, Matthies L, Simoes E, Keilmann L, Hartkopf AD, Sokolov AN, Walter CB, Sickenberger N, Wallwiener S, Feisst M, Gass P, Fasching PA, Lux MP, Wallwiener D, Taran FA, Rom J, Schneeweiss A, Graf J, Brucker SY. Reliability of an e-PRO Tool of EORTC QLQ-C30 for Measurement of Health-Related Quality of Life in Patients With Breast Cancer: Prospective Randomized Trial. J Med Internet Res. 2017 Sep 14;19(9):e322. doi: 10.2196/jmir.8210. PMID 28912116
- See also: Related Info — http://www.jmir.org/2017/9/e322/